CLINICAL TRIAL: NCT03638752
Title: The Impact of Comprehensive Education Before Gastroscopy on Improving the Tolerance of Patients: A Prospective Randomized Controlled Study
Brief Title: The Impact of Comprehensive Education Before Gastroscopy on Improving the Tolerance of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018-R010
Record Dates: First submitted 2018-08-08; First posted 2018-08-20 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Comprehensive Education

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The endoscopist and endoscopy nurse will not know to which treatment arm the patient belongs as only the research assistant will has taken down this information. This information does not travel with the patient to the endoscopy room. The patient is also instructed to not reveal to the endoscopist or endoscopy nurse if he or she has taken or not taken the comprehensive education.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive education group (Experimental): The details of Comprehensive education are as follows:
  1. introduce the purpose, method and function of breathing training and the whole process of gastroscopy;
  2. instruct patients to take deep breath training, inhaling with his/her nose and exhaling with his/her mouth,
  3. provide patients with a disposable dental biting device and repeat exercising deep breathing again until he/she is fully mastered,
  4. inform patients to cooperate with the instructions issued by endoscopist and endoscopy nurse during the whole process of gastroscopy,
  5. inform patients to inhale with nose and exhale with mouth when the gastroscope passes through the throat, then he/she should perform inhaling and exhaling with his/her nose until the end of the gastroscopy when the endoscopist ask to adjust the breathing method,
  6. inform patients that there would be some normal physiological reaction when gastroscopy, such as throat discomfort and nausea/vomiting.
  Interventions: Other: Comprehensive education group
- standard education (No Intervention): The details of standard education are as follows:
  1. inform patients to cooperate with the instructions issued by endoscopist and endoscopy nurse during the whole process of gastroscopy,
  2. inform patients that there would be some normal physiological reaction when gastroscopy, such as the throat discomfort and nausea/vomiting.

INTERVENTIONS:
Other: Comprehensive education group — The details of Comprehensive education are as follows:
  1. introduce the purpose, method and function of breathing training and the whole process of gastroscopy;
  2. instruct patients to take deep breath training, inhaling with his/her nose and exhaling with his/her mouth,
  3. provide patients with a disposable dental biting device and repeat exercising deep breathing again until he/she is fully mastered,
  4. inform patients to cooperate with the instructions issued by endoscopist and endoscopy nurse during the whole process of gastroscopy,
  5. inform patients to inhale with nose and exhale with mouth when the gastroscope passes through the throat, then he/she should perform inhaling and exhaling with his/her nose until the end of the gastroscopy when the endoscopist ask to adjust the breathing method,
  6. inform patients that there would be some normal physiological reaction when gastroscopy, such as throat discomfort and nausea/vomiting.
  Arms: Comprehensive education group

SUMMARY:
This clinical trial is being conducted to assess whether the comprehensive education before gastroscopy could reduce the adverse reactions, such as nausea, vomiting and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 years undergoing routine gastroscopy
2. Informed consent

Exclusion Criteria:

1. Serious coronary heart disease and myocardial injury with serious heart failure
2. Stenosis of the esophagus or cardia obstruction
3. Acute pharyngitis and tonsillitis
4. Acute upper gastrointestinal bleeding
5. Hemodynamically unstable
6. allergy to topical lidocaine
7. Patients did not cooperate or spirit was not normal
8. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Adverse reaction times in gastroscopy | 1 day
  research assistant records nausea/vomiting/retching times in the whole process of gastroscopy

SECONDARY OUTCOMES:
Patients' tolerance scores | 1 day
  At the end of the procedure, the patients were asked about the tolerance in the process of gastroscopy by using a 100-mm visual analogue scale. Tolerance includes the extent of pain and nausea. The endpoints were assigned "no nausea or no pain " to the left and "worst possible nausea or worst pain imaginable " to the right.

OTHER OUTCOMES:
Endoscopists' assessment scores | 1 day
  At the end of the procedure, Endoscopists scored the level of difficulty in introduction of the gastroscope on a 100-mm visual analogue scale. The endpoints were assigned " easiest" to the left and " worst difficult " to the right.
  Endoscopists' satisfaction was assessed with 100-mm VAS for the performances of the endoscopes. The endpoints were assigned " worst dissatisfied" to the left and " Most satisfied " to the right.
Systolic/diastolic blood pressure (SBP/DBP) | 1 day
  Patients were monitored the Systolic/diastolic blood pressure (SBP/DBP) throughout using an electronic multifunctional patient monitor unit. The research assistant records Systolic/diastolic blood pressure (SBP/DBP) on 5 min prior to endoscopic intubation, during endoscopy and at time of entry into the stomach body
Pulse rate (PR) | 1 day
  Patients were monitored the pulse rate (PR) throughout using an electronic multifunctional patient monitor unit. The research assistant records pulse rate (PR) on 5 min prior to endoscopic intubation, during endoscopy and at time of entry into the stomach body.
Oxygen saturation by pulse oximetry (SpO2) | 1 day
  Patients were monitored the Oxygen saturation by pulse oximetry (SpO2) throughout using an electronic multifunctional patient monitor unit. The research assistant records oxygen saturation by pulse oximetry (SpO2) on 5 min prior to endoscopic intubation, during endoscopy and at time of entry into the stomach body.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, PHD, Principal Investigator — Department of Gastroenterology, Ningbo No. 1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided